CLINICAL TRIAL: NCT07172984
Title: The Value of Standardized Respiratory Rate Monitoring Exercises During Rheumatological Infiltration Procedures - A Single-blind, Randomized, Controlled Non-inferiority Study
Brief Title: The Value of Standardized Respiratory Rate Monitoring Exercises During Rheumatological Injection Procedures
Acronym: Respi-IR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Collaborators: Université Savoie Mont Blanc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHMS25001; 2025-A00019-40 (Other: RCB)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Rheumatological Injection; Pain Management; Respiratory Monitoring
Keywords: rheumatological injection; local anesthesia during intra-articular injection; respiratory rate monitoring
MeSH Terms: conditions — Agnosia | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anesthesia group (Active Comparator): Receives local anesthesia with 5 cc of lidocaine before the infiltration procedure.
  Interventions: Procedure: Anesthesia
- breathing group (Experimental): Explanations for performing 5-minute breathing cycles that facilitate the achievement of cardiac coherence, with visual feedback.
  Interventions: Procedure: breathing group

INTERVENTIONS:
Procedure: Anesthesia — Receives local anesthesia with 5 cc of lidocaine before the infiltration procedure.The patient will receive breathing instructions as part of "SHAM" treatment, which will not allow them to achieve cardiac coherence.
  Arms: Anesthesia group
Procedure: breathing group — The procedure will use 5 cc of saline solution instead of the usual anesthesia. Explanations for performing 5-minute breathing cycles that facilitate the achievement of cardiac coherence, with visual feedback.
  Arms: breathing group

SUMMARY:
The goal of this clinical trial is to demonstrate the non-inferiority of standardized breathing control exercises on perceived pain during rheumatological injections procedures compared to standard care consisting of the addition of a local anesthetic. The study population will consist of patients scheduled to undergo therapeutic ultrasound-guided joint or periarticular injection. The main question it aims to answer is:

* Non-inferiority of breathing exercises compared to the addition of local anesthetic on pain and anxiety experienced during an infiltration procedure.
* Correlation between the reduction in pain and anxiety experienced during a procedure and the cardiac coherence score obtained.

Researchers will compare the anesthesia group (Arm A), which will receive local anesthesia with 5 cc of lidocaine before the infiltration procedure to the breathing group (Arm B), which will receive instructions before the injection procedure on how to perform 5-minute breathing cycles to facilitate the achievement of cardiac coherence to see if the pain perceived in Arm B is not greater than the pain perceived in Arm A.

Participants will be kept blind to their randomization group. Arm A (anesthesia) will receive SHAM breathing exercises, while Arm B (breathing) will receive a placebo injection of anesthetic.

DETAILED DESCRIPTION:
This randomized, controlled, single-blind, single-center non-inferiority study aims to evaluate the impact of local anesthesia and breathing exercises on pain and anxiety management during joint or periarticular injections. Participants are patients referred to a rheumatology consultation or referred by an outside physician for injections requiring local anesthesia, such as those performed on the shoulder, elbow, knee, hip, or ankle.

Patients will be kept blind to their randomization group. In both groups, continuous heart rate recording will be performed during the procedure using the EmWave PRO device (to assess cardiorespiratory variability and calculate a cardiac coherence score).

In the "anesthesia" group, local anesthesia with 5 cc of lidocaine will be administered before the infiltration procedure, and the patient will receive breathing instructions as part of "SHAM" management, which will prevent them from achieving cardiac coherence.

In the "breathing" group, patients will perform 5-minute breathing exercises before the procedure (10-second cycles: 5 seconds of inhalation and 5 seconds of exhalation) to enable them to achieve the expected analgesic cardiac coherence. The practitioner performing the procedure will use 5 cc of saline solution instead of the usual anesthesia.

After infiltration, participants' pain, anxiety, and satisfaction will be measured using EVA scale.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo therapeutic ultrasound-guided joint or periarticular injection.
* Patient able to sign an informed consent form to participate in the study

Exclusion Criteria:

* Patient able to sign an informed consent form to participate in the study - - Allergy to the injection product or anesthetic.
* Injection not allowing the use of a local anesthetic due to insufficient joint volume (e.g., fingers/toes).
* Epidural injection via the sacrococcygeal hiatus.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2028-09-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain during rheumatological injection | during injection
  Pain perceived during rheumatological injection measured using the Visual Analog Scale between 0 to 10 (the higher score mean the worst outcome) and compared between groups.

SECONDARY OUTCOMES:
anxiety during procedure | during the procedure
  Anxiety experienced during the procedure, measured by the Visual Analog Scale between 0 to 10, the higher score mean the worst outcome and compared between groups.
Cardiac coherence score | during procedure
  Cardiac coherence score during injection (0 to 100, the higher score mean the better outcome) , provided by the EMWAVE device, compared between the breathing group and the anesthesia group.
pain correlated with cardiac coherence score | end of intervention
  Pain measured using the Visual Analog Scale ( 0 to 10, the higher score mean the worst outcome) , correlated within the experimental group with the cardiac coherence score.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Métropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: No